CLINICAL TRIAL: NCT01134497
Title: A Randomised Phase II Study of Carboplatin With or Without the Addition of the ETAR Inhibitor ZD4054 as Treatment for Patients With Metastatic Breast Cancer
Brief Title: Carboplatin With or Without ZD4054 in Patients With Metastatic Breast Cancer
Acronym: PLANET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: New information on IMP affected the cost/benefit ratio
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPON-804-10; 2010-018837-23 (EudraCT Number)
Record Dates: First submitted 2010-05-27; First posted 2010-06-02 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (control): carboplatin + placebo (Active Comparator): The control arm will consist of up to 6 cycles of carboplatin (AUC5 q21d for 6 cycles) iv over 30 minutes on day 1, plus placebo by mouth on days 1-21 of a 21 day cycle.
  Interventions: Drug: Placebo
- Arm B: carboplatin + ZD4054 (Experimental): The experimental arm will consist of up to 6 cycles of carboplatin (AUC5 q21d for 6 cycles) iv over 30 minutes on day 1, plus ZD4054 (10mg daily) od by mouth on days 1-21 of a 21 day cycle.
  Interventions: Drug: ZD4054

INTERVENTIONS:
Drug: Placebo — The control arm will consist of up to 6 cycles of carboplatin (AUC5 q21d for 6 cycles) iv over 30 minutes on day 1, plus placebo by mouth on days 1-21 of a 21 day cycle
  Arms: Arm A (control): carboplatin + placebo
Drug: ZD4054 — The experimental arm will consist of up to 6 cycles of carboplatin (AUC5 q21d for 6 cycles) iv over 30 minutes on day 1, plus ZD4054 (10mg daily) od by mouth on days 1-21 of a 21 day cycle.
  Other Names: Zibotentan
  Arms: Arm B: carboplatin + ZD4054

SUMMARY:
In this "randomised Phase II trial" all patients will receive carboplatin, with half randomly selected to receive ZD4054. The other half to also receive a dummy pill or placebo, this is so that we can accurately assess how much extra benefit ZD4054 may give. The trial will recruit 132 patients with metastatic breast cancer from across the UK and assess whether adding ZD4054 to carboplatin delays progression of their disease. It will also show whether the side effects of adding ZD4054 to carboplatin chemotherapy are acceptable.

Because ZD4054 has not previously been given with carboplatin to this population, in Stage 1 of the study 6 patients will receive ZD4054 with carboplatin. If there are no untoward side effects with carboplatin and ZD4054 then the trial will proceed to Stage 2 and a further 126 patients will be randomised to receive carboplatin with either ZD4054 or the placebo; neither the patient nor their doctor will know whether she is receiving ZD4054 or placebo.

DETAILED DESCRIPTION:
In the UK about 41,000 patients are diagnosed with breast cancer each year. More and more patients are surviving breast cancer, mostly due to the earlier detection and improvements in treatment. Nevertheless, in about 6% of patients the cancer has already spread to other parts of the body when they are first diagnosed; in a further 30% of patients the cancer comes back elsewhere in their body after initial treatment. Once it has spread to other parts of the body, breast cancer is incurable, with patients living, on average, a further 24 months. The aims when treating patients with metastatic breast cancer are to prolong and improve their day to day life. A number of different chemotherapy drugs are available for treatment of metastatic breast cancer. There is, however, still a need to develop new treatments. The aim of this trial is to use a new drug called ZD4054 combined with an established chemotherapy drug (carboplatin) to see whether this prolongs the period for which patients live with the cancer kept under control.

ZD4054 is a new, oral drug which may help to slow down cancer growth. It works by blocking growth that is controlled by specific proteins on cancer cells called endothelins.

Endothelins act by binding to their endothelin receptors, presence of these receptors have been found in about 45% of breast cancer cases. ZD4054 is an endothelin receptor blocker. We hope to show that adding this new drug increases the effectiveness of carboplatin. We know from trials in other cancers that similar drugs may be able to slow down the growth of tumours.

Metastatic breast cancer (MBC) remains incurable and there has been little change in long term outcomes. Chemotherapy is used to improve symptoms and prolong survival in patients with advanced breast cancer. Nevertheless, most tumours inevitably progress and the clinical response rates to subsequent chemotherapy agents are disappointing. There is, therefore, a need for continued clinical research into new strategies to enhance the effectiveness of currently available chemotherapy agents to improve survival.

The endothelin pathway has been implicated in a number of oncogenic pathways. ET-1 and ETAR are frequently over-expressed in breast cancers and are prognostic for poor outcome. Inhibition of the endothelin pathway enhances cytotoxicity when combined with chemotherapy agents such as carboplatin in pre-clinical models. ZD4054 is a specific inhibitor of ETAR and represents a novel therapeutic target in breast cancer.

This study investigates whether ZD4054, an oral endothelin A receptor (ETAR) inhibitor, in combination with carboplatin chemotherapy, has sufficient activity to warrant a future Phase III trial in patients with advanced/metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* Histological or cytological diagnosis of metastatic breast cancer, or previous histological diagnosis of breast cancer and evidence of metastatic or locally advanced disease unsuitable for local therapy
* No more than 2 prior lines of chemotherapy treatment for metastatic breast cancer
* Life expectancy greater than 12 weeks
* Patients must have previously received or be ineligible for a taxane
* Informed written consent
* Adequate bone marrow and hepatic function
* Haemoglobin ≥ 9.0 g/dl (if no prior transfusion or transfusion more than 4 weeks previously) or ≥ 10.0 g/dl (transfusion within last 4 weeks), absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥100 x 109/L
* Total bilirubin < 1.5 x upper normal limit
* AST and ALT ≤ 2.5 x upper normal limit (or ≤ 5x UNL in the presence of liver metastases)
* Adequate renal function
* GFR ≥ 60 mls/min calculated using Wright Formula or measured by EDTA plasma clearance At least one measurable lesion on CT scanning. Disease measurable by other RECIST v1.1 compatible imaging (e.g. MRI, CXR) or clinically measurable will be allowed as long as the same assessment method is used throughout the trial
* ECOG performance status ≤ 2

Exclusion Criteria:

* Previous treatment with platinum based chemotherapy
* Known brain or leptomeningeal metastases
* Any co-existing medical conditions that, in the Investigator's judgement, may substantially increase the risk associated with the patient's participation in the study or potentially hamper compliance with the study protocol and follow-up schedule
* Concomitant medication unsuitable for combination with trial medication
* Concomitant administration of potent CYP3A inhibitors, specifically: Protease inhibitors (atanazavir, indinavir, nelfinavir, ritonavir, saquinavir), Macrolide antibiotics (clarithromycin, telithromycin), Azole antifungals (ketoconazole, itraconazole, voriconazole), nefazodone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2011-08-16 (Estimated); Study Completion 2011-08-16 (Actual)

PRIMARY OUTCOMES:
PFS (time to event) | 18 weeks of treatment
  PFS (time to event) based on Response Evaluation Criteria in Solid Tumours (RECIST v1.1). Time from enrolment to any progression and/or death. Those progression-free and alive will be censored at time of last follow-up visit.

SECONDARY OUTCOMES:
Safety | 52 weeks
  Safety will be assesssed throughout the trial treatment and during follow-up.
Tolerability | 52 weeks
  Side effects/tolerability will be assesssed throughout the trial treatment and during follow-up. Participants will have the option of continuing ZD4054 even after the 18 week treatment period has been completed. This will be at the discretion of the consultant.
Feasibility | 18 weeks
  The trial will also assess number of participants requiring dose delays or reductions and / or treatment withdrawal

CONTACTS AND LOCATIONS:
Locations (1):
- Wales Cancer Trials Unit, Cardiff, United Kingdom